CLINICAL TRIAL: NCT02789020
Title: Image Parkinson's Disease Progression Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB201600537-N; R01NS052318 (NIH)
Record Dates: First submitted 2016-05-20; First posted 2016-06-02 (Estimated); Results first posted 2023-09-06 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-08

CONDITIONS: Parkinson's Disease
Keywords: Rasagiline
MeSH Terms: conditions — Parkinson Disease | interventions — rasagiline; Magnetic Resonance Imaging

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Rasagiline (Experimental): This group will receive a 1 mg rasagiline tablet to be taken once daily for one year. In addition, the following test will be performed: a Magnetic Resonance Imaging (MRI), functional Magnetic Resonance Imaging (fMRI), the Montreal Cognitive Assessment, Stroop, Digit Span, Hopkins Verbal Learning Test, Brief Test of Attention, Beck Depression Index, Hamilton Anxiety and Depression Rating Scales, Physical Function Performance Test, and Epworth Sleepiness Scale.
  Interventions: Drug: Rasagiline; Device: Magnetic Resonance Imaging; Device: functional Magnetic Resonance Imaging; Other: Physical Function Performance Test
- Placebo (Placebo Comparator): This group will receive a placebo tablet in the same forum as the rasagiline tablet to be taken once daily for one year. In addition, the following test will be performed: a Magnetic Resonance Imaging (MRI), functional Magnetic Resonance Imaging (fMRI), the Montreal Cognitive Assessment, Stroop, Digit Span, Hopkins Verbal Learning Test, Brief Test of Attention, Beck Depression Index, Hamilton Anxiety and Depression Rating Scales, Physical Function Performance Test, and Epworth Sleepiness Scale.
  Interventions: Other: Placebo; Device: Magnetic Resonance Imaging; Device: functional Magnetic Resonance Imaging; Other: Physical Function Performance Test

INTERVENTIONS:
Drug: Rasagiline — Rasagiline will be taken for one year at the dose of 1mg a day. and subjects will undergo functional and structural brain imaging to determine if rasagiline is slowing the progression of Parkinson's Disease in the brain.
  Other Names: Azilect; MAO-B inhibitor
  Arms: Rasagiline
Other: Placebo — A placebo tablet will be taken for one year, once a day, and at the same dose of 1mg. subjects will undergo functional and structural brain imaging to be compared with the group taking the rasagiline intervention.
  Arms: Placebo
Device: Magnetic Resonance Imaging — This test will be performed at baseline and one year.
  Other Names: MRI
Device: functional Magnetic Resonance Imaging — This test will be performed at baseline and one year.
  Other Names: fMRI
Other: Physical Function Performance Test — This test will be performed at baseline and one year.

SUMMARY:
Parkinson's disease (PD) is a neurodegenerative brain disorder that impairs the ability to perform functions such as grooming, dressing, cooking, and other activities of daily living. PD affected between 4.1 and 4.6 million people worldwide in 2005, and it is projected that up to 9.3 million people will be affected by 2030. Although current pharmacological therapies provide beneficial effects on motor symptoms of the disease (tremor, rigidity, and bradykinesia), intolerable disability eventually develops in most patients. A disease-modifying therapy that slows disease progression is a major unmet medical need in PD. Numerous agents have neuroprotective effects in pre-clinical laboratory models, but none have been shown to have indisputable disease-modifying effects in clinical trials for patients with PD.

The purpose of this research study is to investigate how the brain and motor behavior changes in PD over time in response to rasagiline which is a monoamine oxidase-B(MAO-B) inhibitor. The drug rasagiline will be tested in this study as the MAO-B inhibitor. Rasagiline has been prescribed for many years to treat symptomatic Parkinson's disease. It is FDA approved for the treatment of Parkinson's disease but has not been shown to slow disease progression. The outcome and impact of this study will provide the first evaluation of MAO-B inhibitors at slowing the progression of the nigrostriatal pathway using advanced Magnetic Resonance Imaging (MRI) and functional Magnetic Resonance Imaging (fMRI) methods in PD.

DETAILED DESCRIPTION:
Participants will receive baseline testing to confirm a diagnosis of Parkinsonism and to determine eligibility in the research study. Half of the participants in this study will be in a group that will receive the study drug (rasagiline), and half will be in a group that will receive a placebo. A placebo is a pill that is made to look like the study drug, but it does not contain any active ingredients. A computer algorithm will randomly decide group assignment (like the flip of a coin). The study drug will be provided at the end of the first visit. The participants will not know which study drug is received, placebo or rasagiline.

During the research study the following test may occur: (1) questionnaires about quality of life and depression; (2) tests to measure strength and motor function; (3) tests to measure cognition; (4) orientation session to learn a precision gripping task; (5) functional MRI scan of the brain; (6) structural MRI scan of the brain.

ELIGIBILITY:
Inclusion Criteria:

* 96 patients with clinically diagnosed PD. For the PD diagnosis, we will use the University of Kentucky PD brain bank diagnostic criteria implemented by a movement disorders trained neurologist. Only early stage PD within 5 years of diagnosis who have never taken rasagiline will be included. 5 years since diagnosis was chosen to focus on early stages of PD, where MAO-B inhibitors have shown the most promise. PD are eligible to participate if they are age 40-77, Hoehn and Yahr stage < or equal to 2 when on medication, and able and willing to sign informed consent to be randomized to the placebo or active drug arm.

Exclusion Criteria:

* As necessitated by the risks of Magnetic Resonance Imaging, patients who have any type of implanted electrical device (such as a cardiac pacemaker or a neurostimulator), or a certain type of metallic clip in their body (i.e., an aneurysm clip in the brain), are not eligible for participation in the MRI portion of the study.
* Individuals who are claustrophobic will also be excluded from participation.
* Women who are or might be pregnant and nursing mothers are not eligible. Pregnancy tests will be carried out for each female subject prior to the MRI scan.
* Individuals with psychiatric disorders or dementia will be excluded, along with other neurologic and orthopedic problems that impair hand movements and walking.
* Individuals who have a history metalworking involving cutting processes such as grinding, filing, shaving, and threading, will need radiological clearance to participate in this study. Specifically, individuals who report a history of metalworking will be referred to Radiology at Shands University of Florida(UF) for an orbitofrontal x-ray. In addition, individuals who have sustained an eye injury involving metal will also be referred to Radiology at Shands UF for an orbitofrontal x-ray. Shands at UF will provide a written report stating whether the individual is safe for imaging at 3 Tesla. All expenses related to this procedure will be covered by the PI.
* Patients with a prior stroke or brain tumor are excluded. Patients will be excluded if they are unwilling to comply with the study procedures.

Ages: 40 Years to 77 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2023-05-11 (Actual); Study Completion 2023-05-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David E Vaillancourt, PhD., Principal Investigator — University of Florida
Locations (1):
- Laboratory for Rehabilitation Neuroscience, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be available without any personal identifiers included.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 96 participants diagnosed with PD signed the informed consent document for the study. 6 of these individuals did not complete the study protocol for a variety of reasons: 1 person revealed he had a prior stroke so he was disqualified at the visit, 2 people were excluded due to space restrictions in the MRI, and 3 people withdrew due to claustrophobia related to the MRI. Therefore, out of the 96 people who signed the consent (were enrolled), only 90 peoples' data were included/randomized.
Period: Overall Study
Arm/Group | Rasagiline | Placebo
Started | 45 | 45
Completed | 39 | 40
Not Completed | 6 | 5
Not completed — Withdrawal by Subject | 6 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rasagiline | Placebo | Total
Number analyzed (Participants) | 45 | 45 | 90
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 18 | 21 | 39
  >=65 years | 27 | 24 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.02 (7.77) | 63.44 (8.48) | 64.23 (8.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 13 | 29
  Male | 29 | 32 | 61
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 43 | 43 | 86
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 43 | 43 | 86
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 45 | 45 | 90
Montreal Cognitive Assessment [Mean (Standard Deviation); unit: units on a scale] — The MoCA is out of 30 and higher score indicates better cognitive ability. Scores of 24 or under indicate cognitive impairment. The minimum score is 0 and the maximum score is 30.
  units on a scale | 26.64 (2.17) | 25.82 (2.77) | 26.23 (2.50)
Hamilton Rating Scale for Depression [Mean (Standard Deviation); unit: units on a scale] — The Hamilton Depression Scale is scored out of a total of 52. A higher score indicates the patient experiences more depression; scores about 17 are considered moderate to severe. The minimum score is 0 and the maximum score is 52.
  units on a scale | 5.09 (4.38) | 7.02 (6.02) | 6.06 (5.33)
Hamilton Anxiety Rating Scale [Mean (Standard Deviation); unit: units on a scale] — The Hamilton Anxiety Scales is totaled out of 56. A higher score indicates more anxiety experienced by the patient; scores of 25-30 are considered moderate to severe. The minimum score is 0 and the maximum score is 56.
  units on a scale | 8.53 (8.04) | 10.69 (7.94) | 9.64 (8.02)
Parkinson's Disease Questionnaire (PDQ-39) [Mean (Standard Deviation); unit: units on a scale] — The PDQ-39 is scored out a total of 100. A higher score indicates that the patient experiences more deficits as a result of PD. The minimum score is 0 and the maximum score is 100.
  units on a scale | 18.28 (18.84) | 25.93 (20.36) | 22.19 (19.90)
Movement Disorders Society UPDRS [Mean (Standard Deviation); unit: units on a scale] — The max score of UPDRS is 199. A higher score indicates more deficits as a result of PD. The minimum score is 0 and the maximum score is 199.
  units on a scale | 29.62 (10.87) | 32.76 (12.42) | 31.19 (11.71)

OUTCOME MEASURES:

1. Primary Outcome: Change in Free-water Accumulation in the Substantia Nigra
Description: 12-month study in PD to watch the effect of an Monoamine Oxidase-B inhibitor on the progressive increase of free-water accumulation in the substantia nigra.
  Recently, free-water diffusion MRI analysis using a bi-tensor model was developed to explicitly estimate the contribution of freely diffusing water molecules within the voxel. This free-water measure is expected to increase with atrophy-based neurodegeneration. Since substantia nigra degeneration occurs mostly in the posterior region of the substantia nigra in PD (ie. ventrolateral tier), we tested the hypothesis that free-water would be elevated in the posterior substantia nigra of PD.
Time Frame: Baseline and one-year
Measure: Mean (Standard Deviation); unit: arbitrary units (A.U.s)
Arm/Group | Rasagiline | Placebo
Number analyzed (Participants) | 45 | 45
arbitrary units (A.U.s) | 0.0009 (0.01) | 0.0041 (0.01)

2. Primary Outcome: Change in Blood Oxygen Level-dependent(BOLD) Signal in the Posterior Putamen, M1, and Supplementary Motor Area(SMA).
Description: 12-month study in PD to watch the effect of an MAO-B inhibitor on BOLD signal in the posterior putamen, M1, and SMA.
Time Frame: Baseline and one-year
Population: The values below represent the BOLD signal in SMA.
Measure: Mean (Standard Deviation); unit: arbitrary units (A.U.s)
Arm/Group | Rasagiline | Placebo
Number analyzed (Participants) | 45 | 45
arbitrary units (A.U.s) | -0.054 (0.315) | -0.086 (0.251)

3. Secondary Outcome: Changes in Parkinson's Disease Motor Symptoms and Bradykinesia
Description: Motor testing batteries such as the Purdue Pegboard Test will be administered to measure changes in the progression of the PD motor symptoms and bradykinesia.
Time Frame: Baseline and one-year
Measure: Mean (Standard Deviation); unit: count of pegs
Arm/Group | Rasagiline | Placebo
Number analyzed (Participants) | 45 | 45
count of pegs | 1.04 (3.15) | 0.689 (3.94)

4. Secondary Outcome: Changes Between the Groups on fMRI
Description: Participants will use their hand to squeeze an MRI compatible grip force transducer in the MRI unit.
Time Frame: Changes from baseline to 1 year
Measure: Mean (Standard Deviation); unit: unitless
Arm/Group | Rasagiline | Placebo
Number analyzed (Participants) | 45 | 45
unitless | -0.054 (0.315) | -0.086 (0.251)

ADVERSE EVENTS:
Time Frame: 1 year (the follow-up occurred one year after the baseline visit)
Description: Documented in a running table and submitted to University of Florida Institutional Review Board for acknowledgement
Arm/Group | Rasagiline | Placebo
All-Cause Mortality (participants affected / at risk) | 0/45 | 0/45
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/45
Other Adverse Events (participants affected / at risk) | 12/45 | 9/45
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rasagiline (N=45) | Placebo (N=45)
Orthostatic Hypotension (Vascular disorders) | 1 (1) | 0 (0) — Patient experienced low blood pressure while on medication, but was unsure if medication is the cause.
Weight Loss (Metabolism and nutrition disorders) | 1 (1) | 0 (0) — Patient experienced weight loss while on medication, but is unsure if medication was the cause.
Hypersexuality (Social circumstances) | 1 (1) | 0 (0) — Patient experienced hypersexuality while on medication, but was unsure if medication is the cause.
Headaches (Nervous system disorders) | 1 (1) | 0 (0) — Patient experienced headaches while on medication, but was unsure if medication was the cause.
Falls (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) — Patient experienced falls while on medication/placebo, but was unsure if medication was the cause.
Hair Loss (Endocrine disorders) | 1 (1) | 0 (0) — Patient experienced hair loss while on medication, but was unsure if medication was the cause.
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) — Patient experienced vomiting while on the placebo, but there should be no connection to the placebo.
Joint Pain/Stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) — Patients experienced joint pain/stiffness while on medication/placebo, but was unsure if medication was the cause.
Vertigo/Dizziness (Nervous system disorders) | 0 (0) | 1 (1) — Patient experienced vertigo/dizziness while on placebo, but there should be no connection to the placebo.
Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Patient experienced congestion while on placebo, but there should be no connection to placebo.
Edema (Vascular disorders) | 0 (0) | 1 (1) — Patient experienced edema while on placebo, but there should be no connection to placebo.
Fatigue (Social circumstances) | 1 (1) | 2 (2) — Patients experienced fatigue while on medication/placebo, but was unsure if medication was the cause.
Light-Headedness (Nervous system disorders) | 2 (2) | 1 (1) — Patient experienced light-headedness while on medication/placebo, but was unsure if medication was the cause.
Increased Resting Tremor (Nervous system disorders) | 1 (1) | 0 (0) — Patient experienced increased resting tremor while on medication, but was unsure if medication was the cause.
Dizziness and Light-Headedness (Nervous system disorders) | 1 (1) | 0 (0) — Patient experienced both dizziness and light-headedness while on medication, but was unsure if medication was the cause.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-06-29): https://cdn.clinicaltrials.gov/large-docs/20/NCT02789020/Prot_SAP_000.pdf
  • Informed Consent Form (2020-03-30): https://cdn.clinicaltrials.gov/large-docs/20/NCT02789020/ICF_001.pdf